CLINICAL TRIAL: NCT01795456
Title: Contrast Enhanced Ultrasound for Assessment of Carotid Artery Neovascularization as a Marker of Disease Activity in Takayasu's Arteritis and Giant Cell Arteritis
Brief Title: Carotid Artery Neovascularization in Takayasu's and Giant Cell Arteritis
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-595
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Takayasu's Arteritis; Giant Cell Arteritis; Arteritis; Vasculitis; Aortitis
Keywords: Takayasu's arteritis; Giant Cell arteritis; Arteritis; Vasculitis; Aortitis; Disease Activity; Carotidynia; Neovascularization; Carotid Intima Media Thickness
MeSH Terms: conditions — Takayasu Arteritis; Giant Cell Arteritis; Arteritis; Vasculitis; Aortitis; Neovascularization, Pathologic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the ability of contrast enhanced carotid ultrasound to serve as an indicator of disease activity in patients with Takayasu's arteritis or Giant Cell arteritis and to determine if patients with active arteritis have a thickening of their blood vessel walls compared to healthy people of the same age and gender.

DETAILED DESCRIPTION:
Takayasu's arteritis and Giant Cell arteritis are chronic, relapsing diseases of the large arteries which can lead to significant narrowing of the arteries through episodes of inflammation within the artery walls. The changes in the vessel walls will be determined by an ultrasound test looking at and measuring: carotid vessel wall changes called carotid Intimal-Media Thickness (cIMT) and the presence of new blood vessels (neovascularization) using a contrast agent. Ultrasound findings will be correlated with markers of inflammation in the blood, findings from other radiology studies (such as MRI) already ordered as part of routine clinical care, and physical exam findings and symptoms of consistent with disease activity. 15 arteritis patients and 5 healthy controls will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 years
* Diagnosis of Takayasu's arteritis or giant cell arteritis
* Suspicion of common carotid involvement on the basis of physical examination (cervical bruit), carotidynia, documented CCA involvement on an imaging study (MRA, CTA, or ultrasound), or documented upper extremity large vessel involvement on an imaging study (MRA or CTA or ultrasound).
* Ability to provide informed consent

Exclusion Criteria:

* Prior stroke, carotid surgery or angioplasty
* Pregnant (or trying to become pregnant)
* Nursing
* Known or suspected cardiac shunt
* Documented hypersensitivity to the contrast agent
* Severe pulmonary hypertension or unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, serious ventricular arrhythmias, or respiratory failure)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Takayasu's arteritis or giant cell arteritis will be screened from the clinics of the Vasculitis Clinic and the Vascular Medicine Clinic at the Cleveland Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Correlation between carotid IMT and neovascularization and disease activity | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Soo Hyun Kim, MD, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Section of Vascular Medicine, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No